CLINICAL TRIAL: NCT02809846
Title: Quell Opioid Reduction and Pain Relief in Patients With Cancer
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Unable to recruit enough participants.
Sponsor: Scripps Translational Science Institute (Other)
Collaborators: NeuroMetrix, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: IRB-16-6815
Record Dates: First submitted 2016-06-20; First posted 2016-06-22 (Estimated); Results first posted 2020-01-21 (Actual); Last update posted 2020-01-21 (Actual); Status verified 2019-04

CONDITIONS: Pain; Metastatic Breast Cancer; Prostate Cancer; Colorectal Cancer
MeSH Terms: conditions — Pain; Breast Neoplasms; Prostatic Neoplasms; Colorectal Neoplasms

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Quell Device (Active Comparator): Quell is a class II medical device with FDA 510(k) clearance for the symptomatic relief and management of chronic intractable pain, without a prescription. It operates by using an electrical stimulator to activate peripheral sensory nerves and trigger analgesia.
  Interventions: Device: Quell
- Sham Quell Device (Sham Comparator): Identical to Active Comparator, but provides sub-therapeutic electronic stimulation.
  Interventions: Device: Sham Quell

INTERVENTIONS:
Device: Quell
  Arms: Quell Device
Device: Sham Quell
  Arms: Sham Quell Device

SUMMARY:
To study effects the Quell device has on opioid consumption and pain relief in patients with cancer.

DETAILED DESCRIPTION:
Single site, double blinded, placebo controlled randomized clinical trial. 40 subjects will be selected based on the inclusion criteria and then randomized to either the intervention group or the placebo control group. Prior to the start of this study, a Controlled Substance Utilization Review and Evaluation (CURES) reports will be acquired to establish baseline number of opioid prescriptions for each subject. Subjects will track how consistently they are using pain medications, both opioids and non-opioids, during the two weeks prior to the start of the study. They will also provide twice daily recordings of their pain intensity via a mobile application. At the end of this two-week period, each subject will be fitted with a Quell device or a sham device, including initial calibration to the subject's comfort level as described in the background section.Once the study subjects have started using the device, we will also be able to monitor and track their sleep wirelessly via the mobile application as long as they are wearing the device. Subjects will receive weekly check in's to monitor the functionality of the device and to help troubleshoot any issues with the device for the duration of subject participation in the study. These check-ins will take place in person, by phone, and or per subject's usual outpatient oncology visits. Each subject will use their device for 8 weeks, during which they will continue to track their pain, sleep and frequency of pain medication use as stated above. Study investigators will receive automated alerts via email to ensure that study are participants using their devices and that the devices are powered on at regular intervals for the duration of the study.Total duration of subject participation will be 10 weeks.

ELIGIBILITY:
Inclusion Criteria:

1. Male or Female greater than or equal to 18 year of age at visit one.
2. Documented diagnosis of metastatic breast, prostate or colorectal cancer with a prognosis of 6 month or greater as determined by the primary oncologist.
3. Visual evidence that subject owns a smart phone and is able to use basic mobile applications such as downloading an app, opening the app, and performing one simple task within the app.
4. Subject speaks and reads English fluently.
5. Subject able to understand and grant informed consent.
6. Live in an area with cellular data connectivity available as provided by the subject.
7. Documented adherence with clinic follow up visits per medical records.
8. Subject using at least one opioid medication on a daily basis.

Exclusion Criteria:

1. Subject has a cardiac pacemaker, implanted defibrillator or other implanted electronic device.
2. Inability to complete subjective data as required; e.g. on mobile application and questionnaires.
3. Does not live in an area with suitable cellular data connectivity.
4. Has infrequent scheduled clinic visits.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 33 (Actual)
Dates: Start 2016-07 (Actual); Primary Completion 2017-08 (Actual); Study Completion 2017-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Lase Ajayi, MD, Principal Investigator — Scripps
Locations (1):
- Scripps Translational Science Institute, La Jolla, California, United States

IPD SHARING:
Plan to Share IPD: Undecided

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Study was conducted at the Scripps Mercy Oncology Clinic in San Diego California. Enrollment began on Wednesday 7/5/216. The last participant completed on 7/27/17 . The trial was terminated before reaching the projected sample size because of unanticipated difficulties in the recruitment and retention of individuals with targeted conditions.
Groups:
- Quell Device: Quell is a class II medical device with FDA 510(k) clearance for the symptomatic relief and management of chronic intractable pain, without a prescription. It operates by using an electrical stimulator to activate peripheral sensory nerves and trigger analgesia.
  For the active device, a therapy session consisted of one hour of continuous stimulation with high frequency electric nerve stimulation varying between 60 and 100 Hz.
  Quell
- Sham Quell Device: Identical to Active Comparator, but provides sub-therapeutic electronic stimulation.For the sham device, a therapy session consisted of three 2-minute periods of stimulation at 0, 28 and 58 minutes with a frequency that also varied between 60 and 100 Hz
  Sham Quell
Period: Overall Study
Arm/Group | Quell Device | Sham Quell Device
Started | 17 | 16
Completed | 8 | 9
Not Completed | 9 | 7

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Quell Device | Sham Quell Device | Total
Number analyzed (Participants) | 17 | 16 | 33
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 15 | 13 | 28
  >=65 years | 2 | 3 | 5
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7 | 10 | 17
  Male | 10 | 6 | 16
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 1 | 1
  Black or African American | 4 | 0 | 4
  White | 11 | 14 | 25
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 2 | 1 | 3
Region of Enrollment [Number; unit: participants]
  United States | 17 | 16 | 33

OUTCOME MEASURES:

1. Primary Outcome: Change in Daily Opioid Use Assessed as Recorded by the Subject in Their Analgesia Diary.
Description: The primary end point of this study was the difference in the change in daily opioid use between the active device group and the sham device group, assessed at weeks 2, 4, 6, 8, and 10 of the study as recorded by the subject in their analgesia diary. Participants documented which medication was taken, how much, and at what time. Dose and type of opioid pain medication was converted to morphine milliequivalents (MME) using conversion factors published by the Centers for Medicare and Medicaid Services (CMS)and combined as a daily dose for each day in a subject's analgesia journal.
Time Frame: Weeks: 2,4,6,8,10
Measure: Mean (Standard Deviation); unit: MME
Arm/Group | Quell Device | Sham Quell Device
Number analyzed (Participants) | 8 | 9
MME
  Week 0 (Baseline) | 51.1 (40.8) | 41.3 (46.7)
  Week 10 | 27.0 (33.7) | 38.5 (15.6)
Statistical Analysis 1: Comparison: Quell Device vs Sham Quell Device; Initially, a sample size of 20 participants per treatment group (active and sham) was selected to achieve 90% power to find a 20% difference in mean percent change in opioid consumption between the two groups with an estimated standard deviation of 22% and 80% power to detect the same difference with a standard deviation of 19% at a two-sided alpha = 0.05; Test type: Other — Bivariate associations between variables were assessed using statistical methods appropriate for the variable types. Baseline characteristics (demographics, other morbidities, baseline medication use, pain intensity and QOL) were compared between the two treatment groups to assess effectiveness of randomization and identify important covariates for multivariable analyses. Associations between demographic variables and primary and secondary endpoints were examined; p < 0.05, Mixed Models Analysis — Sensitivity analyses comparing use of data from all participants with use of participants with complete data only was also performed. Agreement between different measures representing the same variable type was assessed using correlation analyses; Multivariable analysis with mixed effect regression models were used to assess the effect of treatment group on the primary and secondary outcomes; Similar models were used to assess associations of treatment group with secondary endpoints. Model fit was assessed by Akaike's Information Criteria to determine optimal covariance structure

ADVERSE EVENTS:
Time Frame: Adverse events were tracked from the moment of enrollment till the subject completed the study or was discontinued from the study.
Arm/Group | Quell Device | Sham Quell Device
All-Cause Mortality (participants affected / at risk) | 1/17 | 0/16
Serious Adverse Events (participants affected / at risk) | 0/17 | 0/16
Other Adverse Events (participants affected / at risk) | 0/17 | 4/16
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Quell Device (N=17) | Sham Quell Device (N=16)
Device sensitivity (Skin and subcutaneous tissue disorders) | 0 (0) | 4 (4) — One subject in the sham device group had increased sensitivity to the device electrodes. These adverse effects did not cause any physical harm, 3 individuals discontinued the study early due to device intolerance.

LIMITATIONS AND CAVEATS:
Recruitment and attrition rates were major limitations of this study.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2016-12-16): https://cdn.clinicaltrials.gov/large-docs/46/NCT02809846/Prot_000.pdf
  • Statistical Analysis Plan (2019-01-17): https://cdn.clinicaltrials.gov/large-docs/46/NCT02809846/SAP_001.pdf